CLINICAL TRIAL: NCT03463291
Title: Role of MRI Diffusion in Differentiation Between Benign and Malignant Bony Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A.M. Attia, principal investigator, Assiut University
Other Study IDs: MRIBMBL
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Efficacy of MRI Diffusion in Differentiation Between Benign and Malignant Bony Lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: All patients with bony lesions
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — * T1 weighted image.
  * Fast spin-echoT2 weighted image.
  * Short inversion recovery (STIR).
  * T1-fat suppressed images.
  * Diffusion weighted sequences with different b values 0-1000 s/mm2 with qualitative assessments by the different b values as well as quantitative assessment by measurement of the ADC values.

SUMMARY:
Bone tumors are categorized according to their tissue of origin into cartilagenous, osteogenic, fibrogenic, fibrohistiocytic, haematopoietic, vascular, and lipogenic tumors.

Magnetic resonance imaging (MRI) is now indispensable for the preoperative workup and therapeutic follow-up of patients with musculoskeletal tumors.

The application of DW-MRI in bone marrow is today an established examination technique that provides a unique contrast and that can help in the detection of bone-marrow pathologies and the differentiation of benign and malignant bone-marrow lesions.

Diffusion MRI provides quantitative and qualitative assessments of tissue cellularity and cell-membrane integrity. It is widely used for tumour detection, characterisation, and monitoring during treatment. Diffusion MRI supplies functional information that complements the structural evaluation.

In combination with standard structural MRI parameters, the ADC value improves tumour characterization. Diffusion MRI can also be used to monitor tumours during chemotherapy. Tumour necrosis results in loss of cell membrane integrity and in expansion of the extracellular compartment, leading to greater water-molecule diffusion with an increase in the ADC value.

ELIGIBILITY:
Inclusion Criteria:

* All patients with bony lesions will be included in the study.

Exclusion Criteria:

* Patient with cardiac pacemaker.
* Patients with metallic prosthesis in the region of examination.
* Patients with claustrophobia.
* Patient with recent history of surgical or imagining guided biopsy from the bony lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited outpatient clinic of Assiut General hospital and Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The ADC value of MRI diffusion in benign and malignant bony lesions ( considering ADC value <1.2 ..malignant while ADC>1.2 ..benign) | 1 day